CLINICAL TRIAL: NCT07236879
Title: Effects of Artificial Intelligence-based Diabetic Retinopathy Screening on Timely Access to Treatment in Individuals With Diabetes
Brief Title: Artificial Intelligence for Diagnosing Diabetic Retinopathy in Primary Care
Acronym: AID-DR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); TelessaúdeRS / UFRGS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 2024-0238
Record Dates: First submitted 2025-06-04; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Retinopathy
Keywords: screening; diabetic retinopathy; artificial intelligence
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: The AID-DR trial is designed as a randomized, controlled, double-blinded, non-inferiority trial with two parallel groups and a primary endpoint of adequate referrals to specialized care. Randomization will be performed in a 1:1 ratio using variable block sizes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RDIA group (Experimental): The proposed intervention is the provision of universal screening for DR with retinography performed on a mobile fundus camera under mydriasis supported by a computer program in adults with diabetes mellitus; based on the diagnosis made by the computer program, patients will be classified as having referable DR or not, and referral to a specialist will be based on this classification.
  Interventions: Diagnostic Test: Mobile retinography interpreted by artificial intelligence
- RDOF group (Active Comparator): The proposed control is the provision of universal screening for DR in adults with diabetes mellitus with retinography performed on a mobile fundus camera under mydriasis and with obtained images being interpreted remotely by ophthalmologists; based on the diagnosis made by the ophthalmologist, patients will be classified as having referable DR or not, and referral to a specialist will be based on this classification.
  Interventions: Diagnostic Test: Mobile retinography interpreted by ophthalmologists

INTERVENTIONS:
Diagnostic Test: Mobile retinography interpreted by artificial intelligence — All participants will undergo mobile retinal photography in primary care by a trained nursing assistant. If randomized to RDIA group, their photos will be analyzed by artificial intelligence.
  Arms: RDIA group
Diagnostic Test: Mobile retinography interpreted by ophthalmologists — All participants will undergo mobile retinal photography in primary care by a trained nursing assistant. If randomized to RDOF group, their photos will be interpreted remotely by ophthalmologists.
  Arms: RDOF group

SUMMARY:
This is a clinical trial to evaluate the effects of universal screening for diabetic retinopathy (DR) and diabetic macular edema (DME) using artificial intelligence (AI) in the interpretation of fundus photographs obtained by trained nursing assistant using a portable fundus camera in a primary care setting, compared with images obtained by the same method, but interpreted by ophthalmologists.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years old) diagnosed with diabetes mellitus who agree to participate in the study.

Exclusion Criteria:

* Any contraindication for pharmacological mydriasis (such as knowledge of having closed-angle glaucoma, pregnancy).
* Life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 922 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of appropriate referrals to ophthalmologist | Through study completion, an average of 1 year
  Appropriate referrals: asymptomatic patients with moderate to severe nonproliferative DR, proliferative DR, significant macular edema, and uninterpretable exams. This data will be obtained by reviewing the medical records of ophthalmological in-person consults of included patients.

SECONDARY OUTCOMES:
Number of patients referred for laser sessions | Through study completion, an average of 1 year
  Considering only patients referred for argon laser sessions aiming retinal photocoagulation for the treatment of diabetic retinopathy. This data will be obtained through access to the medical records of patients referred for specialized care.
Number of pharmacological intraocular treatment | Through study completion, an average of 1 year
  Considering treatment with anti-VEGF drugs or intravitreal corticosteroids for the treatment of diabetic retinopathy and diabetic macular edema. This data will be obtained through access to the medical records of patients referred for specialized care.
Referral failure | After study completion, an average of 15 months
  Screening with false negative result. This data will be obtained by an independent ophthalmologist review of all images of the not referred patients.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz D Schaan, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chagas TA, Dos Reis MA, Leivas G, Santos LP, Gossenheimer AN, Melo GB, Malerbi FK, Schaan BD. Prevalence of diabetic retinopathy in Brazil: a systematic review with meta-analysis. Diabetol Metab Syndr. 2023 Mar 2;15(1):34. doi: 10.1186/s13098-023-01003-2. PMID 36864478
- [Background] Schneiders J, Telo GH, Lavinsky D, Dos Reis MA, Correa BG, Schaan BD. Organizational intervention to improve access to retinopathy screening for patients with diabetes mellitus: health care service improvement project in a tertiary public hospital. Prim Care Diabetes. 2023 Aug;17(4):354-358. doi: 10.1016/j.pcd.2023.05.007. Epub 2023 Jun 14. PMID 37328386
- [Background] Dos Reis MA, Kunas CA, da Silva Araujo T, Schneiders J, de Azevedo PB, Nakayama LF, Rados DRV, Umpierre RN, Berwanger O, Lavinsky D, Malerbi FK, Navaux POA, Schaan BD. Advancing healthcare with artificial intelligence: diagnostic accuracy of machine learning algorithm in diagnosis of diabetic retinopathy in the Brazilian population. Diabetol Metab Syndr. 2024 Aug 29;16(1):209. doi: 10.1186/s13098-024-01447-0. PMID 39210394